CLINICAL TRIAL: NCT05991349
Title: A Phase 1/2 Study of IBI129 in Subjects With Unresectable, Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of IBI129 in Subjects With Unresectable, Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI129A101
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI129 (Experimental): IBI129
  Interventions: Drug: IBI129

INTERVENTIONS:
Drug: IBI129 — Subjects will receive IBI129 on Day 1 of a 21-day cycle (or intervals determined by the Investigator and Sponsor based on safety, toxicity and PK data), until unacceptable toxicity, disease progression, withdrawal of consent, occurrence of other reasons for discontinuing study therapy, or for a maximum of 24 months of treatment, whichever occurs first.

SUMMARY:
This is a phase 1/2 multicenter, first-in-human study of IBI129. It includes a phase 1 dose escalation and expansion section to identify MTD/RP2D of IBI129, plan to enroll 22~180 subjects, and a phase 2 to explore efficacy, safety and tolerability of IBI129 at RP2D in specified types of solid tumor. Approximately 182 evaluable subjects will be enrolled for phase 2

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol;
2. At least 1 evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.;
3. Male or female subjects ≥ 18 years old;
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1;
5. Anticipated life expectancy of ≥ 12 weeks;
6. Adequate bone marrow and organ function

Exclusion Criteria:

1. Participate in any other interventional clinical research except observational (non-interventional) study or in the follow-up phase of the interventional study;
2. Received previous anti-tumor therapy within 4 weeks or 5 half-lives of the anti-tumor regimens before the first administration of study drug, whichever is shorter.
3. Progressed refractory to an antibody drug conjugate that consists of an exatecan derivative that is a topoisomerase I inhibitor.
4. Plan to receive other antitumor therapy during the study excluding palliative radiotherapy for the purpose of symptom (like pain) relief that must also do not have impact on tumor assessment throughout the study;
5. Known symptomatic central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 24 months
  Occurrence and severity of adverse events (AEs), with severity determined by NCI CTCAE v5.0 criteria
Number of subjects with clinically significant changes in physical examination results | 24 months
  Clinically significant abnormal physical examination findings reported by the investigator.
Number of subjects with clinically significant changes in vital signs | 24 months
  Vital signs including body temperature, pulse, respiratory rate, SpO2 and blood pressure
MTD or RP2D of IBI129 | 12 months
  Number of subjects with dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Plasma concentration (Cmax) of IBI129 | 12 months
  Plasma concentration of IBI129 for single and multiple doses.
Area under the curve (AUC) of IBI129 | 12 months
  AUC of IBI129 for single and multiple doses.
Time to maximum concentration (Tmax) of IBI129 | 12 months
  Tmax of IBI129 for single and multiple doses.
Clearance (CL) of IBI129 | 12 months
  Clearance of IBI129 from the plasma
Volume of distribution (V) of IBI129 | 12 months
  Apparent volume of distribution of IBI129.
Half-life (T1/2) of IBI129 | 12 months
  T1/2 of IBI129 for single and multiple doses.
Immunogenicity of IBI129 | 12 months
  Incidence of anti-drug (IBI129) antibody
Objective response rate (ORR) | 24 months
  ORR as evaluated per the RECIST v1.1 criteria
Duration of response (DoR) | 24 months
  DoR as evaluated per the RECIST v1.1 criteria
Disease control rate (DCR) | 24 months
  DCR as evaluated per the RECIST v1.1 criteria
Time to response (TTR) | 24 months
  TTR as evaluated per the RECIST v1.1 criteria
Progression free survival (PFS) | 24 months
  PFS as evaluated per the RECIST v1.1 criteria
Overall survival (OS) | 24 months
  Overall survival.

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St George private Hospital, Kogarah, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
- China (4):
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - Tianjin Medical university cancer institute & Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No